CLINICAL TRIAL: NCT00507858
Title: A Phase I Dose Escalation Study of Pemetrexed in Patients With Advanced Head and Neck Squamous Cell Cancer
Brief Title: Pemetrexed (Alimta) in Patients With Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0082
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Squamous Cell Cancer; Alimta; Pemetrexed; Dexamethasone; HNSCC; Decadron
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Pemetrexed; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pemetrexed (Experimental): Starting dose 500 mg/m^2 IV once every 3 weeks
  Interventions: Drug: Pemetrexed
- Pemetrexed + IV Dexamethasone (Experimental): Pemetrexed Starting dose 500 mg/m^2 IV once every 3 weeks + Dexamethasone 20 mg intravenous (IV) Day 1.
  Interventions: Drug: Pemetrexed; Drug: Dexamethasone
- Pemetrexed + Oral Dexamethasone (Experimental): Pemetrexed starting dose 500 mg/m^2 IV once every 3 weeks + Dexamethasone 4 mg orally twice daily for 3 Days.
  Interventions: Drug: Pemetrexed; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pemetrexed — Starting dose of 500 mg/m^2 IV Once Over 10 Minutes Every 3 Weeks
  Other Names: Alimta; LY231514; MTA; Multitargeted Antifolate; NSC-698037
Drug: Dexamethasone — Arm 2 = 20 mg IV On Day 1; Arm 3 = 4 mg oral (PO) Twice Daily for 3 Days
  Other Names: Decadron
  Arms: Pemetrexed + IV Dexamethasone; Pemetrexed + Oral Dexamethasone

SUMMARY:
Primary Objective:

* To determine the maximum tolerated doses (MTDs) of pemetrexed when given with dexamethasone. (Please note: One of the three treatment groups will not receive dexamethasone)

Secondary Objectives:

* To assess dose limiting toxicity (DLT), which is defined as grade 4 neutropenia > 7 days duration, neutropenic fever, grade 4 thrombocytopenia, or any grade 3 or 4 non-hematologic toxicity excluding nausea/vomiting and excluding grade 3 transaminase toxicity.
* To determine objective response rate, as defined as complete response (CR) or partial response (PR), confirmed by 2 CT scans at least 6 weeks apart in patients treated with pemetrexed as a single agent with advanced squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
Pemetrexed is designed to block enzymes in the body that are important for tumor growth.

If you are found to be eligible to take part in this study, you will be assigned to one of 3 groups. All participants will receive pemetrexed once every 3 weeks through a needle in the vein over about 10 minutes. Every 3 weeks is considered 1 cycle. Participants in Group 1 will receive pemetrexed only. Participants in Group 2 will also receive dexamethasone on Day 1 of each cycle through a needle in the vein. Participants in Group 3 will take dexamethasone by mouth the day before, the day of, and the day after receiving pemetrexed.

Three (3) different dose levels of pemetrexed will be studied. The first group of 6 participants will be treated at Dose Level 1 (lowest of the 3 doses) and evaluated for 3 weeks. If 0 or 1 out of 6 participants experience severe side effects at Dose Level 1, the next group of 6 participants will be treated at Dose Level 2. At any given dose, if greater than 1 out of 6 participants experience severe side effects, then no further participants will receive that dose or a higher dose.

Every 3 weeks (each cycle), you will have a physical exam, including measurement of vital signs (temperature, pulse, breathing rate, and blood pressure) and weight. Blood (about 3-4 teaspoons) will be collected for routine tests. A performance status evaluation (a test looking at the ability to perform everyday activities) and a liver function test will also be done. Your tumor will be evaluated by CT scan and chest x-ray every 2 cycles of study treatment.

While on study, you will be required to take folic acid by mouth every day for 5-7 days before the first dose of pemetrexed and continuing until 3 weeks after your last dose of pemetrexed. You will also receive an injection of vitamin B12 into your muscle 1 to 2 weeks before your first dose of pemetrexed. The vitamin B12 injection will be repeated every 9 weeks until 3 weeks after your last dose of pemetrexed. It is very important that folic acid and vitamin B12 be given to decrease the risk of severe side effects from the pemetrexed.

You may receive up to 6 cycles of treatment. You will be taken off study if the disease gets worse or intolerable side effects occur. When you stop taking study drug on this study, you will have a physical exam, including measurement of vital signs (temperature, pulse, breathing rate, and blood pressure) and weight. Blood (about 3-4 teaspoons) will be collected for routine tests. A performance status evaluation (a test looking at the ability to perform everyday activities) and a liver function test (about 1-2 teaspoons of blood) will also be done.

After completion of 6 cycles of treatment, you will be asked to return to the clinic for follow-up visits every 2-3 months for standard follow-up.

This is an investigational study. The FDA has approved pemetrexed for the treatment of non-small cell lung cancer. However, the FDA has authorized pemetrexed for research only in the patients with HNSCC. Between 40-50 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed metastatic or recurrent head and neck squamous cell carcinoma from the primary lesions and/or lymph nodes of the oral cavity, oropharynx, hypopharynx, or larynx.
2. Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >/= 20 mm with conventional techniques or as >/= 10 mm with spiral CT scan.
3. Patients have received one or more chemotherapy regimens.
4. Age >/= 18 years.
5. Life expectancy of greater than 3 months.
6. No acute intercurrent illness or infection.
7. ECOG performance status </= 2 (Karnofsky >/= 60%)
8. Laboratory parameters: white blood count (WBC) >3,000/mL; Neutrophils >1,500/mL; Hemoglobin >8g/dL; Platelets >100,000/mL; Bilirubin <1.5 times the upper limit of normal (ULN); Serum creatinine: within normal institutional limits; aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) < 3 times institutional ULN if alkaline phosphatase is < ULN, except in known hepatic metastasis, wherein ALT/AST may be </= 5 times ULN
9. Creatinine clearance: The standard Cockcroft and Gault formula or the measured glomerular filtration rate (GFR) using the appropriate radiolabeled method (51-CrEDTA or Tc99m-DTPA) must be used to calculate CrCl for enrollment or dosing. The same method used at baseline should be used throughout the study. No dosage adjustment is needed in patients with CrCl >/= 45 mL/min.
10. Patients with a history of non-melanoma skin cancer, or other malignancies treated 5 years or more prior to the current tumor, from which the patient has remained continually disease-free, are eligible.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Acute intercurrent illness or infection
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
3. Patients who are receiving any other investigational agents
4. Patients who have known brain metastases
5. Patients who have signs or symptoms of acute infection requiring systemic therapy.
6. Patients having a history of non-melanoma skin cancer, or other malignancies, treated less than 5 years or more prior to the current tumor
7. Patients requiring total parental nutrition with lipids.
8. Patients exhibiting confusion, disorientation, or having a history of major psychiatric illness that may impair the understanding of the informed consent.
9. Patients refusing to sign the informed consent.
10. Histology other than squamous cell carcinoma.
11. Inability or unwillingness to take folic acid or vitamin B12 supplementation
12. Inability to take corticosteroids
13. Inability to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (for short-acting NSAIDs) or 8-day period (for long-acting NSAIDs, such as piroxicam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Pemetrexed | 3 weeks
  MTD for pemetrexed within each schedule of dexamethasone is defined as the highest dose level in which less than 2 instances of dose limiting toxicities (DLT) observed out of 6 treated participants.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org